CLINICAL TRIAL: NCT02003560
Title: Accelerated Partial Breast Irradiation After Breast Conserving Surgery for Low-risk Invasive Breast Cancer: 3D Conformal Radiotherapy (3D-CRT) and Intensity Modulated Radiotherapy (IMRT) - Prospective Phase II Study
Brief Title: Accelerated Partial Breast Irradiation With 3D-CRT and IMRT
Acronym: APERT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Csaba Polgár, Professor, National Institute of Oncology, Hungary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIO-APERT_01
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer; Radiation Toxicity; Side Effects
Keywords: breast cancer; breast conserving therapy; accelerated partial breast irradiation; 3D conformal radiotherapy; intensity modulated radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accelerated partial breast irradiation (Experimental): Accelerated partial breast irradiation delivered by 3 dimensional conformal radiotherapy or intensity modulated radiotherapy
  Interventions: Radiation: accelerated partial breast irradiation

INTERVENTIONS:
Radiation: accelerated partial breast irradiation — 9 x 4.1 Gy accelerated partial breast irradiation delivered by 3D-CRT or IMRT over 5 consecutive days, using twice-a-day fractionation.

SUMMARY:
The purpose of this study is to determine in a phase II clinical trial whether accelerated partial breast irradiation after breast conserving surgery using 3 dimensional external beam radiotherapy (3D-CRT) and intensity modulated radiotherapy (IMRT) for low-risk invasive breast cancer patients is safe without causing serious late radiation side-effects.

DETAILED DESCRIPTION:
It is a sequential phase II trial. Eligible patients after breast conserving surgery (BCS) are treated with accelerated partial breast irradiation (APBI) using three-dimensional conformal radiotherapy (3D-CRT) for the first 45 patients or intensity modulated radiotherapy (IMRT) for the second 45 patients.

Primary end-point of the study: late radiation side-effects at 5 years. Early stopping criteria: Not used as primary end-point is late side-effects. Interim analysis: Not planned Secondary end-points: cosmetic results, quality of life, local recurrence-free survival, regional recurrence free survival, distant metastasis free survival, relapse free survival, overall survival, cancer specific survival.

Null-hypothesis for primary end-point: The incidence of severe (>G2) late radiation side-effects after APBI using 3D-CRT or IMRT will not exceed 10%.

Stratification:

* by treatment delivery: 3D-CRT - first 45 patients; IMRT - second 45 patients
* by bra capsize: Capsize A-B; C; and D-D+

Treatment intervention: 9 x 4.1 Gy APBI using 3D-CRT (first 45 patients) or IMRT (second 45 patients) delivered within 5 days, using twice-a-day fractionation.

Clinical target volume (CTV) and Planning target volume (PTV) definition:

CTV = excision cavity + 20 mm minus the actual pathological surgical margin in mm PTV = CTV + 5 mm in each direction

Follow-up:

* ECOG PS, physical examination (inspection and palpation), registration of side-effects (RTOG (Radiation Therapy Oncology Group) EORTC (European Organization for Research and Treatment of Cancer)) early and late radiation morbidity scoring scheme) and cosmetic results (using the Harvard scale) : 7-14 days after RT, than in every 3 months for 2 years, and every 6 months for 5 years.
* Mammography: at 6, 12, 18, 24 months, and annually thereafter
* Quality of life questionnaire (QLQ) (e.g. EORTC (European Organization for Research and Treatment of Cancer) QLQ-30 and Breast (BR)-23) before RT, at 7-14 days after RT, at 3, 6, and 12 months, and annually thereafter
* digital photography: before treatment, at 7-14 days after treatment, and yearly thereafter

ELIGIBILITY:
Inclusion Criteria:

* previous breast conserving surgery within 12 weeks (in case of adjuvant chemotherapy within 28 days after completion of chemotherapy)
* patient age > 40 years
* ECOG performance status: 0-1
* life expectancy >5 years
* invasive ductal, papillary, mucinous, medullary or tubular carcinoma
* unifocal tumor
* pathological tumor size < or = 30 mm
* pathological negative axillary nodal status with axillary dissection or sentinel lymph node biopsy
* surgical clips in the tumor bed
* pathological surgical free margins of at least 2 mm
* written informed consent of patients

Exclusion Criteria:

* Stage III-IV
* multifocal tumor
* extensive intraductal component (EIC)
* ductal or lobular carcinoma in situ (DCIS or LCIS)
* invasive lobular cancer (ILC)
* lymph-vascular invasion (LVI)
* contralateral breast cancer
* history of treatment for previous breast cancer
* lactation or breast feeding women
* Paget-disease of the nipple
* psychiatric disorder
* increased radiosensitivity (e.g. collagen vascular disease)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-12; Primary Completion 2019-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
late radiation side-effect | 5 years
  Late radiation side-effects at 5 years scored by the RTOG (Radiation Therapy Oncology Group) EORTC (European Organization for Research and Treatment of Cancer) late radiation morbidity scoring scheme

SECONDARY OUTCOMES:
cosmetic results | 5 years
  cosmetic results at 5 years measured by the Harvard criteria
local tumor control | 5 years
  Local tumor control defined as reappearance of the tumor in the ipsilateral breast
regional tumor control | 5 years
  regional tumor control at 5 years
overall survival | 5 years
  overall survival at 5 years
disease free survival | 5 years
  disease free survival at 5 years
cancer specific survival | 5 years
  cancer specific survival at 5 years

OTHER OUTCOMES:
quality of life | 5 years
  quality of life measured by the EORTC (European Organization for Research and Treatment of Cancer) QLQ-30 and BR-23 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Polgár, MD, PhD, MSc, Study Chair — National Institute of Oncology; Norbert Mészáros, MD, Principal Investigator — National Institute of Oncology
Locations (1):
- National Institute of Oncology, Budapest, Hungary

REFERENCES:
- [Derived] Mozsa E, Meszaros N, Major T, Frohlich G, Stelczer G, Sulyok Z, Fodor J, Polgar C. Accelerated partial breast irradiation with external beam three-dimensional conformal radiotherapy. Five-year results of a prospective phase II clinical study. Strahlenther Onkol. 2014 May;190(5):444-50. doi: 10.1007/s00066-014-0633-1. Epub 2014 Mar 12. PMID 24619017